CLINICAL TRIAL: NCT01322022
Title: Treatment of Sleep Disturbances in Young Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO09070340; R34MH082882 (NIH)
Record Dates: First submitted 2011-03-22; First posted 2011-03-24 (Estimated); Results first posted 2015-02-02 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-01

CONDITIONS: Autism; Autism Spectrum Disorders
Keywords: Autism; Autism Spectrum Disorders; Sleep Problems; Sleep Disturbances; Interventions
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Parasomnias | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parent Training (Experimental): Behavioral Intervention
  Interventions: Behavioral: ParentTraining
- Parent Education (Active Comparator): 5 Sessions of individual parent education
  Interventions: Other: Parent Education

INTERVENTIONS:
Behavioral: ParentTraining — 5 sessions of individual parent training
  Other Names: Behavioral intervention; Psychoeducational intervention
  Arms: Parent Training
Other: Parent Education — Parent Education to control for time and attention
  Other Names: Control
  Arms: Parent Education

SUMMARY:
This study will compare the efficacy of a behavioral parent training program (PT) aimed specifically at common sleep disturbances compared to parent education (PE) program focusing on general issues related to autism. In a sample of 40 well characterized young children who meet criteria for an autism spectrum disorder (24-72 months), the investigators will test whether the five session PT program is superior to the PE program in decreasing sleep disturbances.

The primary aim of this study is to evaluate the efficacy and feasibility of a PT program for sleep disturbance in young children with autism compared to PE.

To this end, there are two hypothesis:

* Hypothesis 1: After the end of treatment, PT will be significantly more effective than PE in improving parent reports of a) bedtime struggles and resistance; b) sleep latency; c) night wakings; d) morning wakings; and / or e) sleep association problems as measured by the composite sleep index score from the modified Simonds and Parraga Sleep Questionnaire (MSPSQ; Simond & Parraga, 1982; Wiggs & Stores, 1998).
* Hypothesis 2: At the end of treatment, children in the PT group (n=20) will display significantly improved total sleep period as measured by actigraphy in comparison to children in the PE group (n=20).

The secondary aim of this study is to evaluate the impact of participating in PT on child's daytime behavior and functioning and parenting stress compared to PE.

To measure this aim, there are 4 exploratory hypothesis:

* Exploratory Hypothesis 1: Lower Irritability subscales scores will be reported on both parent and teacher / therapist completed Aberrant Behavior Checklist (ABC) for the PT group than the PE group at 4 weeks and 8 weeks
* Exploratory Hypothesis 2: Lower Child Behavior Checklist (CBCL; parent completed) and Caregiver-Teacher Report Form (C-TRF; teacher completed) scores will be reported for the PT group than the PE group at 4 weeks and 8 weeks.
* Exploratory Hypothesis 3: The PT group will have higher scores on the Vineland Adaptive Behavior Scales: 2nd Edition (VABS-II) at 4 weeks and 8 weeks compared to PE group.
* Exploratory Hypothesis 4: Parents receiving PT will report significantly lower scores on the Parenting Stress Index (PSI) at 4 weeks and 8 weeks compared to parents receiving PE.

DETAILED DESCRIPTION:
Autism Spectrum Disorders (Autistic Disorder, Pervasive Developmental Disorder, Asperger Disorder) are severe developmental disorders of early childhood onset affecting as many as 1 in 150 children (Center for Disease Control & Prevention, 2007). They characterized by deficits in social interaction and communication, as well as repetitive behavior and restricted interests (American Psychiatric Association, 2000). Given the severity and the prevalence, autism is a significant public health issue. Recent years have seen both an increase in the prevalence of autism and an improved ability to diagnose the disorder much earlier (Fombonne, 2003). It is during the child's early years when it is generally agreed that intensive interventions are most likely to improve long term prognosis (National Research Council, 2001). While not a core feature of autism, it is widely accepted that a large percentage children with autism spectrum disorders (autism) present with significant sleep issues (Honomichl, Goodlin-Jones, Burnham, Gaylor & Anders, 2002; Johnson, 1996; Wiggs & Stores, 2004). Sleep problems in typically developing children are known to adversely impact daytime functioning, learning acquisition, as well as parenting and family functioning (Dahl, 1996; Ebert & Drake, 2004; Sadeh, Gruber, & Raviv; 2002; Sadeh, Raviv, & Gruber, 2000). For young children with autism whose development is already compromised by a range of deficits, the detrimental impact of sleep disturbances may be even more significant. However, the impact of sleep disturbances on optimal performance in behavioral and education interventions have not been systematically explored.

This study will conduct a randomized clinical trial to evaluate the efficacy of a behavioral parent training program in the amelioration of sleep disturbances in young children with autism. This work will be used to examine the feasibility, acceptability and efficacy of a behavior training program for sleep disturbance in children with autism. It represents a low cost and rapid clinical approach to the problem in this younger age group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with an autism spectrum disorder
* Presence of sleep disturbance

Exclusion Criteria:

* Medical etiology of sleep disturbance

Ages: 24 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2009-12; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia R Johnson, PhD, Principal Investigator — U of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh Autism Cetner, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Parent Training: 5 sessions of individual parent training to address sleep problems in young children with autism
- Parent Education: 5 Sessions of individual parent education on various topics related to autism (definition, diagnosis, development, therapies, etc.)
Period: Overall Study
Arm/Group | Parent Training | Parent Education
Started | 20 | 20
Week 4 | 15 | 18
Completed | 15 | 18
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parent Training | Parent Education | Total
Number analyzed (Participants) | 15 | 18 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 18 | 33
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 3.51 [2 to 6] | 3.6 [2 to 6] | 3.56 [2 to 6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 11 | 15 | 26
Region of Enrollment [Number; unit: participants]
  United States | 15 | 18 | 33

OUTCOME MEASURES:

1. Primary Outcome: Modified Simond & Parraga Sleep Questionnaire (MSPSQ) - Composite Sleep Index
Description: The MSPSQ used by Wiggs and colleagues (Wiggs & Stores, 1996 ; Wiggs & Stores, 1999 : Wiggs & Stores, 2004) was used to assess the child's sleep quality. It was completed by the primary caregiver for both groups at baseline and at weeks 4 and 8. Using Wiggs & Stores earlier-described conventions for determining the Composite Sleep Index (CSI) score, the CSI was calculated by assigning a score to the frequency of the targeted sleep problems: bedtime resistance, night awakening, early awakening, and sleeping in places other than bed. In addition, scores were assigned for the duration of sleep latency and night awakenings. The total CSI score ranged from 0 to 12, with higher scores indicating more severe bedtime and sleep patterns.
Time Frame: Baseline, Week 4, and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent Training | Parent Education
Number analyzed (Participants) | 15 | 18
units on a scale
  Baseline | 6.53 (2.17) | 7.44 (2.60)
  Week 4 | 4.80 (2.68) | 6.83 (2.50)
  Week 8 | 4.47 (2.90) | 6.28 (2.68)

2. Secondary Outcome: Actigraphy - Total Sleep Time
Description: Measure of total time spent asleep using Motionlogger model actigraph by Ambulatory Monitoring, Inc. (www.ambulatory-monitoring.com) and algorithms in associated software.
Time Frame: Baseline, Week 4, Week 8
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Parent Training | Parent Education
Number analyzed (Participants) | 15 | 18
minutes
  Baseline | 455 (73) | 448 (90)
  Week 4 | 444 (94) | 439 (82)
  Week 8 | 460 (60) | 434 (90)

3. Primary Outcome: Actigraphy - Sleep Efficiency
Description: Measure of sleep efficiency defined as the percentage of time sleeping while in bed with lights off
Time Frame: Baseline, Week 4, Week 8
Measure: Mean (Standard Deviation); unit: Percentage of Time Sleeping
Arm/Group | Parent Training | Parent Education
Number analyzed (Participants) | 15 | 18
Percentage of Time Sleeping
  Baseline | 82 (7) | 85 (10)
  Week 4 | 86 (5) | 86 (8)
  Week 8 | 85 (6) | 86 (10)

4. Primary Outcome: Actigraphy - Sleep Latency
Description: Measure of sleep latency defined by the time from lights off to sleep onset.
Time Frame: Baseline, Week 4, Week 8
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Parent Training | Parent Education
Number analyzed (Participants) | 15 | 18
minutes
  Baseline | 35 (31) | 29 (27)
  Week 4 | 36 (20) | 27 (23)
  Week 8 | 33 (26) | 29 (22)

ADVERSE EVENTS:
Arm/Group | Parent Training | Parent Education
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No